CLINICAL TRIAL: NCT00439400
Title: A Double-Masked, Randomized, Placebo-Controlled Study of ALTY-0501 (Doxycycline 0.025% Ophthalmic Solution) for the Treatment of Dry Eye Administered QID for a 56 Day Period Utilizing the Controlled Adverse Environment Model
Brief Title: A Study of ALTY-0501 for the Treatment of Dry Eye Administered 4 Times a Day for a 56 Day Period
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alacrity Biosciences, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 0600419
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: doxycycline
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: doxycycline
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
The objective of this study is to assess the safety and efficacy of doxycycline 0.025% (ALTY-0501) ophthalmic solution for the treatment of dry eye using the Controlled Adverse Environment (CAE) Model.

DETAILED DESCRIPTION:
Dry eye is the most prevalent form of ocular discomfort and irritation. Estimates range up to 20 million people in the US being affected with mild dry eye, and the literature reports that as many as 3.2 million American women suffer from clinically significant dry eye.(Schaumberg et al, 2003). Dry eye can be related to external factors, such as the low humidity of air conditioned offices, winter heating, a dusty or windy outdoor environment, prolonged use of computers, or wearing of contact lenses, as well as to internal factors, such as hormonal imbalance, autoimmune disease, the presence of many widely prescribed systemic medications, anatomical changes or trauma, and aging. Chronic dry eye disease is associated with an immune-based inflammation of the lacrimal glands and the ocular surface. Symptoms result in mildly decreased quality of life at a minimum, and with increasing severity, loss of function and productivity, pain, light sensitivity, and the misery that accompanies significantly impaired vision and decreased quality of life. With the aging population in the United States and other countries of the developed world, and with increasing computer use, dry eye will become more prevalent.

Doxycycline is a well established anti-infective drug, and has been used systemically by ophthalmologists to treat moderate to severe case of blepharitis for years. Recently it has been demonstrated that doxycycline in low, non-antimicrobial concentrations also has powerful anti-proteolytic and anti-inflammatory properties. Anecdotal reports on the use of 0.025% doxycyline eyedrops in human patients with dry eye and/or meibomian gland disease indicate a significant improvement in ocular surface staining and a significant decrease in patient symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older;
* Are able and willing to follow instructions, including participation in study assessments, and can be present for the required study visits for the duration of the study;
* Have a diagnosis of dry eye associated with meibomian gland disease; A fluorescein staining staining score of ≥ 1+ in at least one region of the cornea; Presence of eyelid telangiectasia and/or inspissation or metaplasia of meibomian gland orifices; An ocular dryness score of ≥1+;
* Have a TFBUT ≤ 7 seconds in at least one eye at Visit 1;
* Have a best corrected visual acuity (BCVA) of +0.7 or better assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Visit 1;
* (If female and of childbearing potential) Are not pregnant, nursing, or planning a pregnancy. Women of childbearing potential are required to have a negative urine pregnancy test at the screening and exit visits and agree to use an acceptable method of contraception for the duration of the study;

Exclusion Criteria:

* Have anterior blepharitis, which is deemed clinically significant and/or likely to interfere with study parameters in the opinion of the investigator;
* Are diagnosed with an on-going ocular infection (bacterial, viral, or fungal), or active ocular inflammation (e.g., follicular conjunctivitis);
* Report an ocular discomfort score of 4 in both eyes at time 0 of CAE exposure at Visit 2;
* Wear contact lenses within 1 week of Visit 1 or throughout the course of the study;
* Have contact lens-induced dry eye;
* Have previously had laser in situ keratomileusis (LASIK) surgery;
* Are currently taking any topical ophthalmic prescription or over-the-counter (OTC) solutions, artificial tears, gels or scrubs and cannot discontinue these medications for the duration of the trial;
* Have used Restasis® within 30 days of Visit 1;
* Have used any eye drops within 2 hours of Visit 1;
* Any eye drop containing BAK as a preservative for 1 week prior to study start;
* Have a systemic disease, or uncontrolled medical condition, that in the opinion of the investigator could interfere with study measurements or subject compliance;
* Are currently taking (at Visit 1) any medication known to cause ocular drying that has not been used on a stable dosing regimen for 30 days prior to Visit 1;
* Are currently pregnant, nursing, or planning a pregnancy;
* (For women of childbearing potential) Be unwilling to submit a urine sample for a pregnancy test at Visit 1 and at exit visit;
* Have received another experimental drug or device within 30 days of visit 1.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-02; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Associates, Andover, Massachusetts, United States

REFERENCES:
- See also: Alacrity Biosciences Web page — http://www.alacritybio.com
- See also: Ophthalmic Research Associates web page — http://www.oraclinical.com